CLINICAL TRIAL: NCT04422990
Title: Clinical Evaluation of a Silicone Hydrogel Daily Wear Monthly Replacement Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLY935-C012
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Results first posted 2022-02-24 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Refractive Errors
Keywords: Vision Correction; Contact Lens
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LID018869 (Experimental): Lehfilcon A silicone hydrogel contact lenses worn in both eyes during waking hours only. Lenses will be worn for a total of 3 months, with monthly planned replacement over the course of the study duration. CLEAR CARE will be used for nightly contact lens cleaning and disinfection.
  Interventions: Device: Lehfilcon A contact lenses; Device: CLEAR CARE
- Biofinity (Active Comparator): Comfilcon A silicone hydrogel contact lenses worn in both eyes during waking hours only. Lenses will be worn for a total of 3 months, with monthly planned replacement over the course of the study duration. CLEAR CARE will be used for nightly contact lens cleaning and disinfection.
  Interventions: Device: Comfilcon A contact lenses; Device: CLEAR CARE

INTERVENTIONS:
Device: Lehfilcon A contact lenses — Investigational silicone hydrogel contact lenses
  Other Names: LID018869
  Arms: LID018869
Device: Comfilcon A contact lenses — Commercially available silicone hydrogel contact lenses
  Other Names: CooperVision® BIOFINITY®; Biofinity
  Arms: Biofinity
Device: CLEAR CARE — Hydrogen peroxide-based contact lens cleaning and disinfecting solution

SUMMARY:
The purpose of this clinical study is to evaluate the safety and performance of an investigational soft contact lens compared to a commercially available soft contact lens when worn in a daily wear modality.

DETAILED DESCRIPTION:
Subjects will be expected to attend 4 office visits: Screening/Baseline/Dispense, Week 1 Follow-up, Month 1 Follow-up, and Month 3 Follow-up/Exit. The total expected duration of participation for each subject is approximately 3-4 months in this daily wear clinical study.

ELIGIBILITY:
Key Inclusion Criteria:

* Successful wear of spherical daily wear frequent replacement soft contact lenses for distance correction in both eyes during the past 3 months for a minimum of 5 days per week and 8 hours per day;
* Manifest cylinder equal to or less than 0.75 diopter (D) in each eye;
* Best spectacle corrected visual acuity (using manifest refraction) of 20/20 or better in each eye;
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Wearing habitual contact lenses in an extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment;
* Habitually wearing Biofinity lenses;
* Monovision or multifocal contact lens wearers;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Trial Lead, CDMA Vision Care, Study Director — Alcon Research, LLC
Locations (13):
- United States (13):
  - Alcon Investigative Site, Los Angeles, California
  - Alcon Investigative Site, Novato, California
  - Alcon Investigative Site, Oakland, California
  - Alcon Investigative Site, San Francisco, California
  - Alcon Investigative Site, Orlando, Florida
  - Alcon Investigative Site, West Palm Beach, Florida
  - Alcon Investigative Site, Downers Grove, Illinois
  - Alcon Investigative Site, Louisville, Kentucky
  - Alcon Investigative Site, New York, New York
  - Alcon Investigative Site, Cleveland, Ohio
  - Alcon Investigative Site, Boiling Springs, South Carolina
  - Alcon Investigative Site, Plano, Texas
  - Alcon Investigative Site, Wichita Falls, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 14 sites located in the United States.
Pre-assignment Details: Of the 158 enrolled, 11 subjects were not dispensed study lenses and were exited from the study as screen failures. This reporting group includes all subjects who were dispensed study lenses (147).
Units Other Than Participants: Eyes
Groups:
- Biofinity: Comfilcon A silicone hydrogel contact lenses worn in both eyes during waking hours only. Lenses were worn for a total of 3 months, with monthly planned replacement over the course of the study duration. CLEAR CARE was used for nightly contact lens cleaning and disinfection.
- LID018869: Lehfilcon A silicone hydrogel contact lenses worn in both eyes during waking hours only. Lenses were worn for a total of 3 months, with monthly planned replacement over the course of the study duration. CLEAR CARE was used for nightly contact lens cleaning and disinfection.
Period: Overall Study
Arm/Group | Biofinity | LID018869
Started | 50; 100 Eyes | 97; 194 Eyes
Completed | 47; 94 Eyes | 96; 192 Eyes
Not Completed | 3; 6 Eyes | 1; 2 Eyes
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Travel | 3 | 0

BASELINE CHARACTERISTICS:
Population: Per Protocol (PP): All randomized subjects exposed to any study lenses evaluated in this study with at least one post-baseline (post-dispense) contact lens corrected distance visual acuity (CLCDVA) assessment, minus all data/subjects that met any of the pre-defined critical deviation or evaluability criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Biofinity | LID018869 | Total
Number analyzed (Participants) | 49 | 92 | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (9.7) | 33.1 (10.8) | 33.2 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 61 | 97
  Male | 13 | 31 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 5 | 5
  Not Hispanic or Latino | 49 | 87 | 136
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12 | 20 | 32
  Black or African American | 0 | 1 | 1
  Chinese | 31 | 61 | 92
  Japanese | 1 | 4 | 5
  Korean | 4 | 6 | 10
  Other Asian | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Contact Lens Corrected Distance Visual Acuity (CLCDVA) at Week 1 Follow-Up
Description: Visual acuity (VA) was assessed for each eye individually with study lenses in place using a letter chart. VA was collected in Snellen and converted to logarithm minimum angle of resolution (logMAR). A logMAR value of 0 equates to 20/20 Snellen visual acuity (normal distance eyesight), with lower logMAR values indicating better visual acuity.
Time Frame: Week 1 Follow-Up
Population: PP: A predefined subset of subjects (those with BCVA of 20/20 or better in each eye at baseline/dispense) from another similar completed registration study, CLY935-C010 (NCT04178720) was combined with this study to attain adequate power for the planned hypothesis testing of the primary and secondary endpoints. This included 49 subjects from CLY935-C012 and 39 subjects from CLY935-C010 in the Biofinity group and 92 subjects from CLY935-C012 and 78 subjects from CLY935-C010 in the LID018869 group.
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Biofinity | LID018869
Number analyzed (Participants) | 88 | 170
Number analyzed (eyes) | 176 | 340
logMAR | -0.06 (0.00) | -0.06 (0.00)
Statistical Analysis 1: Comparison: Biofinity vs LID018869; Test type: Non-Inferiority — Noninferiority in mean CLCDVA was declared if the upper confidence limit was less than 0.10 logMAR; Mixed effects repeated measures model — Since a noninferiority hypothesis is being tested, a p-value is not applicable. Confidence limit is being reported and compared to the noninferiority margin; Least squares mean difference = 0.00, 95% CI 2-sided [-0.01 to 0.01] — Least squares mean difference (LID018869 minus Biofinity)

2. Secondary Outcome: Percentage of Subjects Achieving CLCDVA 20/20 or Better in Each Eye at Week 1 Follow-Up
Description: Visual acuity (VA) was assessed for each eye individually with study lenses in place using a letter chart. VA was collected in Snellen, with 20/20 Snellen visual acuity considered normal distance eyesight. Subjects achieving at least 20/20 Snellen in each eye, left and right, contributed to the analysis.
Time Frame: Week 1 Follow-Up
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Units Other Than Participants: eyes
Arm/Group | Biofinity | LID018869
Number analyzed (Participants) | 88 | 170
Number analyzed (eyes) | 176 | 340
percentage of subjects | 98.8 | 97.0
Statistical Analysis 1: Comparison: Biofinity vs LID018869; Test type: Non-Inferiority — Proportion of subjects was used for the statistical analysis. Noninferiority in proportion of subjects achieving CLCDVA 20/20 or better in each eye was declared if the lower confidence limit was greater than -0.10; Generalized linear mixed model — [p-value comment as in outcome 1, analysis 1]; Difference in proportion = -0.01, 95% CI 2-sided [-0.04 to 0.02] — Lens difference (LID018869 minus Biofinity)

ADVERSE EVENTS:
Time Frame: Adverse events (AE's) were collected from time of consent to study exit, approximately 3 months.
Description: AE's were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of participants. The safety analysis set includes all subjects/eyes exposed to any study lenses evaluated in this study. For treatment-emergent safety analyses, subjects/eyes were categorized under the actual study lenses exposed.
Groups:
- Pre-Treatment: Events reported in this group occurred prior to exposure to the study contact lenses
- Biofinity Ocular; Biofinity Non-Ocular: Events reported in this group occurred while exposed to comfilcon A contact lenses
- LID018869 Ocular; LID018869 Non-Ocular: Events reported in this group occurred while exposed to LID018869 contact lenses
Arm/Group | Pre-Treatment | Biofinity Ocular | Biofinity Non-Ocular | LID018869 Ocular | LID018869 Non-Ocular
All-Cause Mortality (participants affected / at risk) | 0/147 | 0/100 | 0/50 | 0/194 | 0/97
Serious Adverse Events (participants affected / at risk) | 0/147 | 0/100 | 0/50 | 0/194 | 0/97
Other Adverse Events (participants affected / at risk) | 0/147 | 0/100 | 0/50 | 0/194 | 0/97

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/90/NCT04422990/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/90/NCT04422990/SAP_001.pdf